CLINICAL TRIAL: NCT04440410
Title: Non-interventional Study to Evaluate Cutaneous and Circulating Inflammatory Biomarkers for a Novel IRAK4-targeted Therapeutic in Hidradenitis Suppurativa and Atopic Dermatitis Patient Samples
Brief Title: Evaluation of Cutaneous and Circulating Inflammatory Biomarkers in Hidradenitis Suppurativa and Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Kymera Therapeutics, Inc. (Industry)
Collaborators: York Dermatology Clinic and Research Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: YDC-2
Record Dates: First submitted 2020-06-01; First posted 2020-06-19 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Hidradenitis Suppurativa; Dermatitis, Atopic
Keywords: IRAK4
MeSH Terms: conditions — Hidradenitis Suppurativa; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples, skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hidradenitis suppurativa: Subjects with active mild, moderate, or severe HS disease using the HS-PGA assessment
- Atopic Dermatitis: Subjects with active moderate or severe AD disease using the PGA assessment

SUMMARY:
This non-intervention study will identify the biomarker profiles in hidradenitis suppurativa (HS) and atopic dermatitis (AD) (as a comparator) that would have the most utility in interventional studies evaluating efficacy during therapeutic intervention. Study data will also be used to correlate cellular/molecular changes in blood (cells and serum), and tissue, with clinical/histopathological phenotypes.

DETAILED DESCRIPTION:
This study is an exploratory correlative study in subjects with HS or AD. Blood samples and skin biopsies will be collected from all subjects and used to assess the following: cutaneous and circulating inflammatory biomarkers and IRAK4 target levels in primary samples, correlations between cutaneous and circulating inflammatory biomarkers and disease severity, effects of IRAK4 degradation on IRAK4 levels and downstream inflammatory biomarkers in ex vivo-treated whole blood from patients.

De-identified routine clinical data that is collected will be correlated with the research findings.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Active HS or AD disease, diagnosed by PI
3. Patients with mild (HS only), moderate, or severe disease using the HS-PGA or PGA assessment.
4. Must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study, and is willing to participate in the study.

Exclusion Criteria:

1. Patient is currently on a biologic or other immunosuppressive treatment for HS or AD.
2. Use of biologic treatment for HS or AD within 3 months or 5 half-lives, whichever is longer
3. Use of non-biologic immunosuppressive treatment (eg. Cyclosporin) in the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active mild, moderate, or severe HS or active moderate or severe AD disease.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Biomarker Identification | Day 1
  Assessment of cutaneous and circulating inflammatory biomarkers and IRAK4 target levels in primary samples
Determination of Biomarker Correlations | Day 1
  Determine correlations between cutaneous and circulating inflammatory biomarkers and disease severity
Examination of IRAK4 Degradation Effects Ex Vivo | Day 1
  Examine effect of IRAK4 degrader on IRAK4 levels and downstream inflammatory biomarkers in ex vivo-treated whole blood from patients

CONTACTS AND LOCATIONS:
Overall Officials: Afsaneh Alavi, MD, Principal Investigator — York Dermatology Clinic and Research Centre
Locations (1):
- York Dermatology Clinic and Research Centre, Richmond Hill, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No